CLINICAL TRIAL: NCT01453010
Title: Self-directed Upper Limb Training Using a SaeboFlex With Acute Stroke Patients: 8 Single Case Reviews
Brief Title: Self-directed Upper Limb Training Using a SaeboFlex in Acute Stroke
Acronym: SaeboFlex
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colchester Hospital University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/H0302/8
Record Dates: First submitted 2011-09-08; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Stroke
Keywords: SaeboFlex; Stroke rehabilitation; Upper Limb Rehabilitation; Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 8 individual case reviews (Experimental): SaeboFlex Self-directed training
  Interventions: Other: Self-directed Upper Limb SaeboFlex Training

INTERVENTIONS:
Other: Self-directed Upper Limb SaeboFlex Training — Participants undergo a 12 week self directed upper limb training programme with the SaeboFlex upper limb orthosis. Training consists of a maximum of 3 x 45 minute sessions a day.
  Participants are closely monitored at least once a week by a saebo-trained therapist.

SUMMARY:
Arm and hand weakness as a result of stroke occurs in approximately 70% of stroke survivors and causes huge loss of function and independence. A wide range of treatment approaches have been developed to improve motor recovery. Despite treatments, such as Constraint Induced Movement Therapy, showing promise, these in large have been have focused on high-intensity and repetitive task-specific practice. Patients with little hand or finger movements however may not be able to participate actively in task specific training.

The SaeboFlex is a dynamic orthosis, with a spring-loaded feature that facilitates opening of the fingers and hand. This allows the patient to grasp and release objects repeatedly, hence enabling participation in repetitive task practice and increasing potential for motor recovery. Despite the SaeboFlex being used successfully in several centers in the country and internationally, research to provide evidence of effectiveness is scarce. As a consequence funding for the SaeboFlex is limited and usually requires patients' to fund their own.

The study aims to explore the potential benefits and feasibility of participating in a Self-directed SaeboFlex training program to allow repetitive task practice in patients early after stroke.

Subjects will undergo a 12-week training program comprising of a maximum of 3 x 45 minute sessions a day. Activities focus on grasping and releasing balls and reaching for targets, wearing the SaeboFlex for the majority of the session. At the end of each session the SaeboFlex is removed and the hand is incorporated into functional tasks as able. Subjects will be set individualized training program by a Saebo-trained therapist. The program will be graded and progressed at a rate that is appropriate to each individual.

The study will measure and follow-up 8 subjects to explore improvements in recovery and functional ability of the upper limb and affect on dependency levels. It will also explore the level of intensity patients early after stroke can tolerate and how they participate in self-directed therapy. All patients will meet the inclusion criteria and be motivated to undergo the specific SaeboFlex self-directed training program. Subjects will record the time and intensity of their training sessions and also their routine upper limb therapy. Patients will be assessed before, during and after the 3 months training. If these cases show promise the study will support the need for large trials including clinical efficacy and dose finding studies.

ELIGIBILITY:
Inclusion criteria:

Subjects will:

* Be either in-patients on Colchester Stroke Unit or,
* Out-patients following an acute stroke admission to Colchester Stroke Unit
* Be adults who have suffered a stroke between 3 and 84 days before recruitment
* Have an anterior circulation stroke - i.e. must have weakness not ataxia
* Have a substantially paretic hand and fingers and meet the criteria for the SaeboFlex orthosis as below
* Have a previously fully functional upper limb (i.e. previous weakness, severe movement disorders, severe Rheumatoid Arthritis )
* Be able to participate in self directed therapy (i.e. no severe visual or cognitive deficits precluding participation task repetitive practice and recording training times)
* Are medically fit to participate in repetitive task practice as determined by the consultant (or GP if out-patient).

Saebo Flex requirements (inclusion criteria)

Subjects must have:

* A minimum of 15 degrees passive wrist extension (fingers must be extended)
* At least 15 degrees active shoulder motion in any plane
* At least 15 degrees elbow flexion
* At least ¼ range of active finger flexion (IP) flexion

Exclusion criteria:

* Patients that are able to open and close his/her hand completely, 10 times keeping the wrist neutral while maintaining his / her maximum shoulder flexion are too good for the Saebo-flex. Other treatment options should be considered.
* Severe joint deformities that could be worsened by using an orthosis, i.e. RA
* Those patients with extremely poor skin integrity which may be cause irritation or skin damage.
* We will not exclude stroke survivors on the basis of age or gender but subjects will need to be motivated for self-directed study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Change from Baseline in upper limb function to 4, 8 and 12 weeks
  Ability to use the paretic upper limb in functional activity. The ARAT is a test of upper limb function with subsections covering grasp, grip, pinch and gross movement. As the SaeboFlex is aimed at achieving grasp and release this measure appears very appropriate. It has good validity and reliability and is widely used in clinical research.
Motricity Index (MI) | Change from Baseline in upper limb voluntary contraction to 4, 8 and 12 weeks
  The Motricity Index (MI) is a clinical measure of the ability to voluntarily contract paretic muscle. It is an ordinal score with six levels of measurement within each of three categories for the upper limb (pinch grip, elbow flexion and shoulder abduction), has been used widely in clinical research, is valid, reliable and sensitive to change after stroke.

SECONDARY OUTCOMES:
Motor Assessment Scale- Upper Limb Section (UL-MAS). | Change from Baseline in upper limb function to 12 weeks
  The UL-MAS covers three upper limb subsets: upper arm function (six), hand movements and advanced hand activities. Each subtest is scored out of 6, with a maximum score of 18. It has quite recently been recommend that the UL-MAS should be scored non-hierarchally, meaning that every item within the subsets should be scored regardless of its place within the hierarchy. The acceptable internal consistency score obtained verifies the validity and reliability of using the UL-MAS as an independent scale.
Visual Analogue Scale | Change from Baseline to 12 weeks
  A Visual Analogue Scales (VAS) is a type of rating scale that is commonly used to measuring an individuals' rating of their own health. A scale from 1 to10 shall be used for a subjective score of how much the subject rates his or her ability to use their arm in functional tasks
Modified Barthel Index (MBI) | Change from Baseline in Independence level to 4, 8 and 12 weeks
  The Modified Barthel Index is used in the stroke pathway on the ward as part of routine practice.
  It is widely used as assessment tools for clinical decision-making and outcome measurement in clinical research. It has good inter-rater reliability. The original Barthel Index was modified to increase sensitivity to change in functional ability and levels of dependence.
Stroke Impact Scale (SIS) | Change from Baseline to 12 weeks
  The Stroke Impact Scale was developed based on feedback from patients and their caregivers. It measures the aspects of stroke recovery which were found to be important to patients and caregivers as well as stroke experts. After intensive psychometric testing the 59 item Stroke Impact Scale Version 3.0 was developed. The 59 questions of the SIS are broken down into eight domains including strength, hand function, mobility, and activities of daily living, emotion, memory, communication and social participation
Berg Balance Test | Change from Baseline in balance to 4, 8 and 12 weeks
  The Berg Balance Scale has been identified as the most commonly used assessment tool across the continuum from acute care to community-based care in stroke rehabilitation. It has been demonstrated to have strong psychometric properties and be sensitive to change. Balance is not directly linked to independence but is a good predictor of mobility levels and risk of falls, and therefore considered an important measure to include.
Questionnaire | 12 weeks
  These will be carried out at the end of the 12 week training period. The interview will include a set list of questions with open ended answers to enable patients to describe how they found the training and whether their expectations were met.
Adverse effects or events monitoring and recording | throughout 12 weeks
  Any complaints of pain, prolonged reduction in function, reduction on soft tissue length, tone or effects on skin integrity are unexpected but will be closely monitored and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stuck, BSc, Principal Investigator — Colchester Hospital University Foundation NHS Trust
Locations (1):
- Colchester Hospital University Foundational NHS Trust, Colchester, Essex, United Kingdom